CLINICAL TRIAL: NCT05589818
Title: A Phase II Study of the Effects of Pembrolizumab on Quality of Life for Patients With Treatment-Naïve, Advanced or Metastatic NSCLC and Poor Performance Status
Brief Title: Pembrolizumab for Advanced NSCLC and PS 2-3
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Deborah Doroshow, Assistant Professor of Medicine, Icahn School of Medicine at Mount Sinai
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY-22-01144
Record Dates: First submitted 2022-09-26; First posted 2022-10-21 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Non-Small Cell Lung Cancer (NSCLC)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — pembrolizumab

STUDY DESIGN:
Intervention Model Description: Phase II, Interventional, Single-Center, Open-Label, Non-Comparative, Single Cohort, Single-Arm, Trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pembrolizumab (Experimental): Patients will be treated with the standard dose of pembrolizumab (200mg IV every 3 weeks) for the first 12 weeks of the study. After week 12 assessments, patients without objective progression of disease are eligible to transition to Q6W dosing of pembrolizumab 400mg IV.
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: Pembrolizumab — Patients will be treated with the standard dose of pembrolizumab for the first 12 weeks of the study. After week 12 assessments, patients without objective progression of disease are eligible to transition to Q6W dosing of pembrolizumab 400mg IV. Patients will be offered this schedule, also an FDA-approved option, at the discretion of the treating physician, based on tolerability of the q3week regimen and clinician assessment of need for closer follow up intervals. Pembrolizumab will be continued until disease progression, unacceptable toxicity, withdrawal of consent, or death.
  Other Names: PD-1

SUMMARY:
This single center open-label trial will enroll a single cohort of patients with advanced non-small cell lung cancer (NSCLC) who are ineligible for treatment with curative intent due to 1) disease stage IV, or 2) inability to tolerate intensive surgery or chemo-radiation. Patients will be eligible for the trial if ISMMS reviewed samples from tumor biopsy have a PDL-1 TPS ≥ 1% and have ECOG performance status rated 2 or 3. All patients will receive anti PD-1 therapy with pembrolizumab 200mg IV every 3 weeks, during which patients will also undergo serial QOL assessments.

This trial will follow a phase II single arm, open label design. The study will enroll 45 patients evaluable for the primary endpoint of which will be change in QOL as measured by the EORTC's QLQ-C30 between Day 1 and Day 84 +/- 7 days. Secondary outcomes including evaluation for development of confounding mental health conditions will be evaluated via serial HADS assessments. Concomitant radiographic assessment with PET/CT, regardless of the doses of pembrolizumab received, will allow for evaluation of secondary efficacy outcomes, including disease response by RECIST 1.1 criteria.

DETAILED DESCRIPTION:
Primary Objective To assess the effects of first-line pembrolizumab upon patient quality of life in patients with metastatic non-small cell lung cancer who are ineligible for standard first line treatments due to poor performance status (ECOG PS of 2 or 3).

Secondary Objectives

* To assess the clinical outcomes of first-line pembrolizumab in this patient population.
* To evaluate the toxicity of first-line pembrolizumab in this patient population.
* To assess patient reported QOL in the emotional domain (using HADS).
* To assess baseline patient-reported performance status and correlate with QOL and clinical outcomes.
* To assess baseline geriatric assessment score for patients 70 years of age and older and correlate with QOL and clinical outcomes.
* To correlate QOL and outcomes with demographic and clinical factors including: age, gender, race/ethnicity, zip code, insurance type, presence/absence of CNS metastases, PD-L1 TPS (<1%, 1-49%, ≥50%), geriatric assessment scores, presence or absence of other major organ dysfunction (e.g. CKD), ECOG 2 vs 3, adverse events: G2, G3-4.

Primary Endpoint Change in QOL score after 12 weeks of treatment as measured by EORTC's QLQ-C30

Secondary Endpoints

* Change in QOL score after 6 weeks of treatment as measured by EORTC's QLQ-C30
* Change in QOL score after 6 and 12 weeks of treatment as measured by EORTC's QLQ-LC13.
* Change in QOL score in the emotional domain after 6 and 12 weeks of treatment as measured by HADS
* Overall survival
* Objective response rate, as determined by independent radiology review and assessed using the Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1, at 12 weeks after treatment
* Progression free survival
* Emergency room visits and hospitalizations
* Adverse events, as assessed by the Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0
* Patient reported ECOG performance status and correlation with QOL and clinical outcomes.
* Treating physician clinical assessment of whether poor PS, as measured by the ECOG Performance Status Scale, is due to disease, other comorbidities, or both and correlation with QOL and clinical outcomes
* Geriatric assessment at baseline for patients 70 years of age and older and correlation with QOL and clinical outcomes, using the Cancer Aging and Research Group (CARG) Chemo-Toxicity Calculator Survey https://www.mycarg.org/?page_id=4480
* Patient Reported Outcome (PRO) completion rate
* Difference in QOL score objective response proportion (CR + PR), and OS at 12 weeks between categories of:

  * Age group
  * Gender
  * Race/ethnicity
  * Zip code
  * Insurance type
  * Presence/absence of CNS metastases
  * PD-L1 (TPS <1%, 1-49%, ≥50%)
  * Geriatric assessment scores
  * Presence or absence of other major organ dysfunction
  * ECOG PS 2 vs 3
  * Adverse events G2, G3-4

Study Drug, Dose, Route, and Regimen: Pembrolizumab 200 mg IV every 3 weeks for 12 weeks, with the option to transition to pembrolizumab 400 mg IV every 6 weeks thereafter. Pembrolizumab will then be continued until disease progression, unacceptable toxicity, withdrawal of consent, or death.

Statistical Considerations: This is a phase II clinical trial to assess the change in Quality of Life (QoL), measured by EORTC QLQ-C30 scores, for patients with treatment-naïve, advanced or metastatic NSCLC and ECOG 2/3 on Pembrolizumab treatment. The global QoL (QLQ-30) at baseline in 218 lung cancer patients had a mean of 57.6 and standard deviation (SD) of 24.3. The research team will test the difference in the change in QoL score between baseline and 12 weeks after Pembrolizumab treatment. A meaningful change, as documented in the literature, has determined to be a 10 score difference. The SD of the change is 18.9, assuming that the pre-/post- correlation is 0.7. A sample of 31 achieves 81% power to detect a mean of paired differences of 10 with an estimated SD of differences of 18.9 and with a significance level of 0.05 using a two-sided paired t-test. Considering the potential 30% drop-out, this study will enroll 45 patients to ensure at least 31 evaluable patients.

Approximately 20 new patients with metastatic NSCLC are seen per month at the Mount Sinai Hospital and Mount Sinai Chelsea sites; of these, approximately 7-8 have a PS of 2-3 based on past experience. Thus, the study can reasonably expect to accrue 2 patients per month to the study, with approximately 24 months needed to complete accrual.

Total number of participants: 45 Estimated Enrollment Period: 24 Months Estimated Duration of Participation: 24 Months Estimated Study Duration: 40 Months Participating Sites: Mount Sinai Hospital and Mount Sinai Chelsea

ELIGIBILITY:
Inclusion Criteria:

* Men and women, aged 18 years and older, with locally advanced NSCLC who are ineligible for definitive surgical resection or concurrent chemoradiation, or metastatic NSCLC
* Patients must not have received any systemic therapy for metastatic cancer
* Patients must not have received any PD-1 or PD-L1 inhibitor
* ECOG performance status of 2 or 3 at the time of consent and on the first day of therapy
* Patients may not have a molecular alteration in ALK, ROS1, EGFR, BRAF, NTRK, RET, MET, or any other gene for which first-line FDA approved targeted therapy exists.
* Patients with treated brain metastases are eligible if there is no evidence of progression for at least 4 weeks after CNS-directed treatment, as ascertained by clinical examination and brain imaging (MRI or CT) during the screening period.
* Patients with new or progressive brain metastases (active brain metastases) or leptomeningeal disease are eligible if the treating physician determines that immediate CNS directed therapy is not required and is unlikely to be required during the first cycle of therapy.
* Patients with HIV on effective anti-retroviral therapy with an undetectable viral load within 6 months are eligible for this trial.
* Adequate organ and marrow function as defined below:

  * Leukocytes ≥ 3,000/mcL
  * Absolute neutrophil count ≥ 1,000/mcL
  * Platelets ≥ 100,000/mcl
  * Total bilirubin ≤ 1.5 x ULN
  * AST (SGOT)/ALT (SPGT) ≤ 3 x ULN or ≤5 x ULN if liver metastases present
  * GFR (Cockroft-Gault) ≥ 30 mL/min
* Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test within 3 days prior to C1D1 of pembrolizumab therapy. For the purposes of this trial, WOCBP are defined as women who have had a menstrual period within the last 48 months.
* Provision of signed and dated informed consent form
* Ability to take the study medication, and complete the study questionnaires
* Stated willingness to comply with all study procedures for the duration of the study
* For women of reproductive potential, agreement to use highly effective contraception during study treatment and for at least 4 months after the final dose
* For men of reproductive potential, agreement to use condoms or other methods to ensure effective contraception with female partners of reproductive potential

Exclusion Criteria:

* Autoimmune conditions requiring >10mg prednisone (or its equivalent) of daily therapy or other systemic immunosuppressive therapy.
* Patients who are receiving other investigational agents
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Patients with known leptomeningeal disease for which CNS therapy is required
* Pregnant or lactating patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2023-05-26 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Change in EORTC QLQ-C30 Quality of Life score | Baseline and 12 weeks post-treatment
  Change in quality of life (QOL) score at 12 weeks post-treatment compared to baseline with pembrolizumab as measured by the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30). The scale ranges from 1=very poor to 7 = excellent. The higher the score the better the quality of life.

SECONDARY OUTCOMES:
Change in EORTC QLQ-C30 Quality of Life score | Baseline and 6 weeks post-treatment
  Change in Quality of Life (QOL) score at 6 weeks post-treatment compared to baseline with pembrolizumab as measured by the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30). The scale ranges from 1=very poor to 7 = excellent. The higher the score the better the quality of life.
Change in EORTC's QLQ-LC13 Quality of Life (QOL) score | Baseline and 6 weeks post-treatment
  Change in Quality of Life (QOL) score at 6 weeks post-treatment compared to baseline with pembrolizumab as measured by EORTC's QLQ-LC13.
  The EORTC QLQ-LC13 is a disease-specific 13-item self-administered questionnaire for lung cancer, to be used in conjunction with the EORTC QLQ-C30. It comprises both multi-item and single-item measures of lung cancer-associated symptoms (ie, coughing, hemoptysis, dyspnea, and pain) and side effects from conventional chemotherapy and radiotherapy (ie, hair loss, neuropathy, sore mouth, and dysphagia). Scores from 0 to 100 were derived for each symptom item, with higher scores representing greater level of symptoms.
Change in EORTC's QLQ-LC13 Quality of Life (QOL) score | Baseline and 12 weeks post-treatment
  Change in Quality of Life (QOL) score at 12 weeks post-treatment with pembrolizumab as measured by EORTC's QLQ-LC13.
  The EORTC QLQ-LC13 is a disease-specific 13-item self-administered questionnaire for lung cancer, to be used in conjunction with the EORTC QLQ-C30. It comprises both multi-item and single-item measures of lung cancer-associated symptoms (ie, coughing, hemoptysis, dyspnea, and pain) and side effects from conventional chemotherapy and radiotherapy (ie, hair loss, neuropathy, sore mouth, and dysphagia). Scores from 0 to 100 were derived for each symptom item, with higher scores representing greater level of symptoms.
Change in Hospital Anxiety and Depression Scale (HADS) Quality of Life (QOL) score | Baseline and 6 weeks post-treatment
  Change in Quality of Life (QOL) score at 6 weeks post-treatment in the emotional domain as measured by HADS. HADS is 14-items scale with responses scored from 0-3, scores for each subscale from 0 (normal) to 21 (severe symptoms). Scores for the entire scale is 0 to 42, with higher score indicating more distress.
Change in Hospital Anxiety and Depression Scale (HADS) Quality of Life (QOL) score | Baseline and 12 weeks post-treatment
  Change in Quality of Life (QOL) score at 12 weeks post-treatment in the emotional domain as measured by HADS. HADS is 14-items scale with responses scored from 0-3, scores for each subscale from 0 (normal) to 21 (severe symptoms). Scores for the entire scale is 0 to 42, with higher score indicating more distress.
Overall Survival (OS) | at 12 weeks post-treatment
  Overall Survival (OS) is defined as the time from the first dose of study treatment to the date of death (whatever the cause).
Objective Response Rate | at 12 weeks post-treatment
  Objective response rate, as determined by independent radiology review and assessed using the Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1:
  Complete Response (CR) Disappearance of all target lesions for a period of at least one month.
  Partial Response (PR) At least a 30% decrease in the sum of the longest diameter of measures lesions (target lesions), taking as reference the baseline sum of the longest diameter.
  Stable Disease (NR/SD) Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum of the longest diameter since the treatment started.
  Progressive Disease (PD) A 20% or greater increase in the sum of the longest diameter of measured lesions (target lesions), taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions
Progression-Free Survival (PFS) | at 12 weeks post-treatment
  Progression-Free Survival (PFS) is defined as the duration of time from start of treatment to the first occurrence of disease progression or death on study from any cause, whichever occurs earlier
Number of Emergency Room Visits | at 12 weeks post-treatment
  Number of Emergency Room Visits
Number of Hospitalizations | at 12 weeks post-treatment
  Number of Hospitalizations
Number of Adverse Events | at 12 weeks post-treatment
  Number of Adverse events, as assessed by the Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0
Patient Reported Eastern Cooperative Oncology Group (ECOG) performance status | at 12 weeks post-treatment
  Patient reported Eastern Cooperative Oncology Group (ECOG) performance status (PS). The ECOG measures level of functioning in terms of daily living abilities:
  0-Fully active, able to carry on all pre-disease performance without restriction
  1. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, eg.light house work
  2. Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about >50% of waking hours
  3. Capable of only limited selfcare; confined to bed or chair >50% of waking hours
  4. Completely disabled; cannot carry on any selfcare; totally confined to bed or chair
  5. Dead
Physician reported ECOG Performance Status Scale | at 12 weeks post-treatment
  Treating physician clinical assessment of performance status, as measured by the ECOG Performance Status Scale
  The ECOG performance status scales and criteria are used by doctors and researchers to assess how a participant's disease is progressing, how the disease affects the daily living, and determines appropriate treatment and prognosis. Grade 0, fully active, able to carry on all pre-disease performance without restriction. Grade 1, restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work. Grade 2, ambulatory and capable of all selfcare, but unable to carry out any work activities; up and about more than 50% of waking hours. Grade 3, capable of only limited selfcare; confined to bed or chair more than 50% of waking hours. Grade 4, capable of only limited selfcare; confined to bed or chair more than 50% of waking hours.
Cancer Aging and Research Group (CARG) Chemo-Toxicity Calculator Survey Score | Baseline
  Geriatric assessment at baseline for patients 70 years of age and older, using the Cancer Aging and Research Group (CARG) Chemo-Toxicity Calculator Survey https://www.mycarg.org/?page_id=4480. CARG scores can range from 0 to 19, with a higher score indicating higher risk of chemotherapy toxicity. CARG scores from 0 to 5 are considered low risk, 6 to 9 are considered intermediate risk, and 10 to 19 are considered high risk.
Patient Reported Outcome (PRO) completion rate | at 12 weeks post-treatment
  PRO completion rate as measured by the percentage of survey instrument questions answered

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Doroshow, MD, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai; Bailey Fitzgerald, MD, Study Director — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 3 months and ending 5 years following article publication.
Access Criteria: Researchers who provide a methodologically sound proposal. To achieve aims in the approved proposal. Proposals may be submitted up to 36 months following article publication. After 36 months the data will be available in our University's data warehouse but without investigator support other than deposited metadata. Information regarding submitting proposals and accessing data may be found at (Link to be included in the URL field below).